CLINICAL TRIAL: NCT00671268
Title: Multicentre, Multinational Randomised DBPC Clinical Trial for Evaluation of Safety and Efficacy of Specific Immunotherapy With Recombinant Major Allergens of Timothy Grass Pollen Adsorbed Onto Aluminium-hydroxide in Patients With IgE-mediated Allergic Rhinoconjunctivitis +/- Controlled Asthma
Brief Title: Evaluation of Safety and Efficacy of Specific Immunotherapy With Recombinant Major Allergens of Timothy Grass Pollen Adsorbed Onto Aluminium-hydroxide in Patients With IgE-mediated Allergic Rhinoconjunctivitis +/- Controlled Asthma
Acronym: AMETHYST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL0704rP; 2007-003208-37 (EudraCT Number)
Record Dates: First submitted 2008-04-23; First posted 2008-05-05 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Rhinoconjunctivitis
Keywords: Grass pollen allergy; specific immunotherapy
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): strict subcutaneous
  Interventions: Biological: AL0704rP
- 2 (Placebo Comparator): strict subcutaneous
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AL0704rP — strict subcutaneous
  Other Names: "na"
  Arms: 1
Biological: Placebo — strict subcutaneous
  Other Names: "na"
  Arms: 2

SUMMARY:
Efficacy and Safety from a high-dosed subcutaneous recombinant preparation

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinoconjunctivitis attributable to grass pollen
* Positive SPT
* Positive EAST
* Positive provocation test

Exclusion Criteria:

* serious disease
* other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2008-03; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change of Symptom and Medication score | during the baseline and the following two pollen seasons

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Professor, Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-003208-37/DE